CLINICAL TRIAL: NCT00182299
Title: A Randomized Clinical Trial Comparing the Effectiveness of Rotator Cuff Repair With or Without Augmentation With Porcine Small Intestine Submucosa (SIS) for Large Rotator Cuff Tears: Pilot Study Phase
Brief Title: An RCT to Compare the Outcomes of Patients With Large Rotator Cuff Repair That Undergo Repair With or Without SIS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); DePuy Orthopaedics (Industry); London Health Sciences Centre (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 63140-1
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: porcine small intestine submucosa (SIS)

SUMMARY:
The prognosis for patients with large rotator cuff tears is poor. This recently developed biologic scaffold provides numerous structural and functional properties that may direct cell growth and aid in tendon healing. To date, there are no randomized clinical trials assessing the effectiveness of the patch to augment repairs of large rotator cuff tears. We propose a study to compare the rate of repair failure, quality of life, function, pain, and range of motion in 60 patients with large rotator cuff. Patients will be randomized (like flipping a coin) to undergo a standard rotator cuff repair with or without augmentation with SIS. Patients are assessed at 6 weeks, 3, 6, 12, 18, and 24 months post-operative

DETAILED DESCRIPTION:
Objective of the full randomized trial To compare the effectiveness of a standardized method of rotator cuff repair with or without augmentation using porcine small intestine submucosa (SIS) in patients with large rotator cuff tears.

Objectives of the pilot study

1. To obtain a preliminary estimate of the likely success of SIS.
2. To formally evaluate our ability to successfully recruit eligible patients into this study.
3. To determine appropriate length of follow up through examination of the pattern of incremental improvement and stabilization of quality of life over time following rotator cuff repair.
4. To determine a more accurate estimation of sample size for the full trial using quality of life.
5. To determine the frequency with which surgeons comply with the surgical protocol.
6. To determine the frequency with which patients and physiotherapists comply with the suggested physiotherapy protocol.

ELIGIBILITY:
Inclusion Criteria:

Patients with large rotator cuff tears (Type 1B or Type 2) determined by clinical examination and diagnostic imaging. Criteria described by Harryman et al (1991) will guide the classification of rotator cuff tears defined and reassessed at the time of surgery (Type 0 = intact cuff, Type 1A = thinned cuff or partial thickness defect, Type 1B= full thickness defect on one tendon, Type 2 = full thickness defect of two tendons, Type 3 = full thickness defect of three tendons).

Exclusion Criteria:

* Previous shoulder surgery, excluding acromioplasty or diagnostic arthroscopy.
* Inability of the surgeon to repair the tear with remaining defect no greater than 10mm in diameter,
* Inability of the surgeon to repair the tear with less than 1cm of medialization,
* Evidence of other significant shoulder pathology including, Type II-IV SLAP lesion, Bankart lesion, Hill Sachs lesion, Grade III osteoarthritis).
* Active joint or systemic infection,
* Significant muscle paralysis of the shoulder girdle,
* Major medical illness that would preclude undergoing surgery,
* Patients who are unwilling or unable to be assessed according to study protocol for one year following surgery
* Major psychiatric illness, developmental handicap or inability to read and understand the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
MRI defined failure of the cuff repair at 2 years postoperative

SECONDARY OUTCOMES:
Quality of life (WORC, ASES), function (SST, CONSTANT), general health (SF-36), pain (VAS), analgesic use; forward flexion; internal/external rotation; lateral elevation

CONTACTS AND LOCATIONS:
Overall Officials: Dianne M Bryant, PhD, Principal Investigator — Western University, Canada
Locations (1):
- The University of Western Ontario, London, Ontario, Canada